CLINICAL TRIAL: NCT01358500
Title: An Assessment of Fentanyl Dose Requirements in Opioid-maintained Individuals
Acronym: FEN001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Adelaide (Other)
Responsible Party: Principal Investigator, Prof Paul Rolan, Professor, University of Adelaide
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEN001
Record Dates: First submitted 2011-05-20; First posted 2011-05-23 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Opioid Dependence
Keywords: opioid dependence; tolerant; dependent
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fentanyl (Experimental)
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — Intravenous infusion using STANPUMP

SUMMARY:
This study seeks to determine the suitable doses of fentanyl with acceptable adverse effect and safety profile in opioid-dependent patients. The investigators anticipate that a well tolerated dose of fentanyl which produces demonstrable analgesia will be found and will be related to the patient's maintenance opioid dose.

DETAILED DESCRIPTION:
Fentanyl is a synthetic opiate with a (clinical) potency of 50 to 100 times that of morphine. Because of its high lipid solubility, fentanyl has a rapid onset of action and a relatively short duration of action. Fentanyl is one of the most widely used agents in the synthetic opioids family. Being a pure agonist with no active metabolites, it is highly suitable for use in patients with opioid tolerance. It can be used outside of an intensive-care clinical environment.

Evidence-based guidelines for clinicians on which agents to use, what doses should be considered and whether treatment doses are related to the dose and the pharmacological properties of the maintenance opioid are lacking, but needed. This study seeks to determine the suitable doses of fentanyl required in opioid-tolerant patients, which are able to overcome the tolerance and hyperalgesia while maintaining an acceptable therapeutic index. The importance of this study is that it has the potential to improve acute pain management in the opioid-tolerant population.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 to 65.
2. Maintained on any opioid with oral morphine equivalent daily dose (MEDD) of 60 mg and above.
3. Have adequate intravenous access for drug infusion.
4. Are currently abstaining from oral and intravenous recreational drug use.

Exclusion Criteria:

1. Known positive for Hepatitis B, Hepatitis C or HIV
2. Contraindication to cold pain testing e.g. cardiac or vascular disease especially Raynaud's phenomenon, blood pressure problems, diabetes, epilepsy and recent serious injury.
3. Using medication which affects pupil size e.g. glaucoma
4. Visual acuity poorer than 6 / 25 corrected (so that saccadic eye movements can be performed correctly.
5. Patients with respiratory insufficiency and poor respiratory drive. The criteria will be a spirometry reading of less than 70% the predicted value and/or having resting oxygen saturation levels of less than 95% on air.
6. Subject is pregnant and/or lactating.
7. Chronic use of benzodiazepines which cannot be withheld for 5 half-lives of the benzodiazepine the patient is on.
8. Known intolerance to fentanyl or other opioids
9. Patients taking tramadol.
10. Patients taking CYP3A4 inhibitors like amiodarone, azole antifungals, cimetidine, clarithromycin, cyclosporine, diltiazem, erythromycin, fluoroquinolones, grapefruit juice, HIV protease inhibitors, metronidazole, quinine, selective serotonin reuptake inhibitors (SSRIs) and tacrolimus.
11. A positive urine test for benzodiazepines on the day of screening or testing.
12. A positive breathalyzer test on the day of testing.
13. Creatinine clearance < 30ml/min as estimated by Cockcroft-Gault formula.
14. Patients with bradyarrythmia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-03 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Attainment of analgesia | Within 2 hours after starting the infusion
  Attainment of analgesia as evidenced by having the cold pain tolerance test reading to twice the baseline value or reaching the absolute value of 2 minutes.

SECONDARY OUTCOMES:
Pupillometry | Within 2 hours after infusion starts
  The pupil diameter will be measured every 30 minutes during the infusion.
Saccadic eye movement | Within 2 hours after infusion starts
  The average peak velocity of the saccadic eye movement will be measured every half an hour for 2 hours.
Morphine Benzedrine Group Scale | Within 2 hours after infusion starts
  This paper test will take 3 minutes to complete and will measure the degree of euphoria.
Electroencephalography (EEG) | Within 2 hours after infusion starts
  The delta, theta and alpha Fz-Cz and Pz-Oz activity will be measured every 30 minutes during the infusion.
Subjective Opioid Withdrawal Scale | Within 1 hour after infusion stops
  This paper test will take 3 minutes to complete and will measure the degree of withdrawal. It will be done at 15, 30 and 60 minutes post infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Rolan, MD, Principal Investigator — University of Adelaide
Locations (1):
- PARC, Royal Adelaide Hospital, Adelaide, South Australia, Australia

REFERENCES:
- [Background] Lotsch J. Pharmacokinetic-pharmacodynamic modeling of opioids. J Pain Symptom Manage. 2005 May;29(5 Suppl):S90-103. doi: 10.1016/j.jpainsymman.2005.01.012. PMID 15907650
- [Background] Mitra S, Sinatra RS. Perioperative management of acute pain in the opioid-dependent patient. Anesthesiology. 2004 Jul;101(1):212-27. doi: 10.1097/00000542-200407000-00032. No abstract available. PMID 15220793